CLINICAL TRIAL: NCT02477904
Title: Ketogenic Diet Therapy for Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: University of Hawaii (Other)
Responsible Party: Principal Investigator, Ryan Lee, MD, Director - Neurodevelopmental Clinic, Research, Shriners Hospitals for Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HON1403
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Autism Spectrum Disorder; Ketogenic Diet; Biochemical Profiles
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ASD/KD (Experimental): Children (2-21 years of age) diagnosed with autism spectrum disorder (ASD) will receive the ketogenic diet (KD) intervention.
  Interventions: Other: Ketogenic Diet
- ASD/non-KD (Active Comparator): Children (2-21 years of age) diagnosed with autism spectrum disorder (ASD) will not receive the ketogenic diet (KD) intervention.
  Interventions: Other: Ketogenic Diet
- non-ASD/non-KD (Active Comparator): Typically developing children (2-21 years of age) diagnosed as not having autism spectrum disorder (ASD) will not receive the ketogenic diet (KD) intervention.
  Interventions: Other: Ketogenic Diet

INTERVENTIONS:
Other: Ketogenic Diet — Dietary
  Other Names: Classic Ketogenic Diet; Shriner's Ketogenic Diet; Non-Ketogenic Diet

SUMMARY:
This study will assess the effectiveness of the ketogenic diet (high-fat, low-carbohydrate, and moderate protein) in treating autism spectrum disorder (ASD). Three study groups will be comprised of children (2-21 years of age) based on whether or not they have ASD and receive the ketogenic diet - ASD/ketogenic diet, ASD/non-ketogenic diet, and non-ASD/non-ketogenic diet.

DETAILED DESCRIPTION:
Recent studies have shown that the ketogenic diet (high-fat, low-carbohydrate, and moderate protein; induce a shift from the primary metabolism of glucose to ketones) or Modified-Atkins diet may be effective in treating autism. Research on the Black and Tan BRachyury (BTBR) T+tf/J mouse strain, characterized by an autism-like behavioral phenotype, has demonstrated the efficacy of a ketogenic diet in improving autism. Although, modified diets, such as the Feingold diet, low-sugar diet, or gluten-free diet, have shown behavioral improvements in patients with Attention Deficit Hyperactivity Disorder (ADHD), the ketogenic diet has not been studied in autism spectrum disorder (ASD) despite the high incidence of ADHD comorbidity. The findings from only one prospective, pilot study have been published, which reported significant behavioral improvement in all 18 autistic subjects after six months (assessed at intervals of four weeks on the diet and two weeks diet-free) on the ketogenic diet. Clearly, the ketogenic and other modified diets as promising treatments for ASD have been understudied. Additional clinical research is necessary to establish the ketogenic diet as a safe, effective treatment alternative for children with ASD.

This proposed research project will involve an ethnically diverse sample (varied genetic background and environmental exposure) to assess the efficacy of the ketogenic diet as a therapeutic intervention, and to understand its beneficial effects in children with ASD. The investigators anticipate that noteworthy findings will contribute to the sparse literature on ASD and effective dietary interventions and prompt future research collaborations with investigators from other medical centers and/or academic institutions. Funding for future research appears promising considering that ketogenic therapies are also a novel method for the treatment of a variety of disorders, including other neurodevelopmental disorders, diabetes, migraine headaches, brain tumors, multiple sclerosis, and obesity.

In addition, the investigators propose to also examine the potential changes in blood composition and intestinal (gut) microbiome in children with (without) ASD who are treated (not treated) with the ketogenic diet in light of the effect on their ASD symptomatology. The relationship between the gastrointestinal tract and the central nervous system has garnered increasing interest in the research community. The gut-brain interface describes a bidirectional relationship in which the central nervous system influences the gut and vice versa. Little is known about the mechanisms behind anecdotal reports of dietary success in humans, but it is suspected that alterations in gut microflora are involved. Mulle et al. (2013) postulated that the connection between the gut microbiome and ASD may be either the direct cause or as indirect consequence of atypical patterns of feeding and nutrition. Similarly, diet patterns, including the ketogenic diet, impact nutrient availability and thus indirectly modulate the gut microbiome. Multiple studies have confirmed differences in levels of gut commensals and overall metabolite profiles in fecal and urinary samples from healthy children compared to children with ASD, potentially as a result of changes in the microbiome. In the maternal immune activation mouse model of ASD, Hsiao et al. (2013) reported that probiotic treatment with B. fragilis could correct behavioral abnormalities and metabolomics profile typified in ASD and ameliorate ASD-relevant GI barrier deficits in mice. Sandler et al. (2000) demonstrated that oral vancomycin treatment showed short-term improvements in children with regressive-onset autism, suggesting that alterations in gut bacteria profile, in this case with antibiotic therapy, may improve autistic behavior. Studies of the gut microbiome in children with ASD may elucidate the role of diet and the alterations in gastrointestinal microbes related to ASD. As a result of these data, novel treatments may be discovered.

The specific aims of this study are:

Aim 1. To evaluate the effect of the ketogenic diet on the core symptoms of autism. The following instruments will be used to measure core autistic symptoms: a) Autism Diagnostic Observation Schedule - Second Edition (ADOS-2); b) Asperger Syndrome Diagnostic Scale (ASDS); c) Childhood Autism Rating Scale (CARS-2); d) Gilliam Autism Rating Scale (GARS-3); e) Social Responsiveness Scale - Second Edition (SRS-2); f) Diagnostic and Statistical Manual IV Text Revision (DSM-IV-TR) and DSM-V ASD criteria; g) Standardized social & intelligence tests (if available, administered by child's school); and h) Vanderbilt ADHD Diagnostic Teacher Rating Scale Forms (Vanderbilt).

Hypothesis: Participants who have ASD/on the ketogenic diet will have significantly lessened core autistic symptoms than those that have ASD/not on the ketogenic diet, between baseline to three and six months after the dietary intervention is initiated.

Aim 2. In anticipation of significant changes in core autistic symptomatology, to examine the effects of the ketogenic diet on the (a) number and dosage of medications used for behavioral management, (b) number of lab tests ordered for behavioral management, (c) number of emergency room or hospital visits for behavioral management, and (d) subject/family satisfaction with the ketogenic diet.

Hypothesis: The number (and/or dosage) of medications, lab tests ordered, and emergency room or hospital visits for behavioral management will decrease, and participant/family satisfaction will be high for participants who have ASD/on the ketogenic diet than those who have ASD/not on the ketogenic diet, between baseline to three and six months after the dietary intervention is initiated.

Aim 3. To compare differences and/or changes in (a) biochemical profiles as defined from blood and stool (gut or fecal microbiome) specimen samples and (b) serum and urine ketone levels.

Hypothesis: Participants who have ASD/on the ketogenic diet will have notably different biochemical profiles and significantly higher serum/urine ketone levels than those who have ASD/not on the ketogenic diet and typically developing controls on a regular diet, between baseline to three and six months after the dietary intervention is initiated.

The investigators anticipate that the KD will be effective in treating ASD, and further an understanding of dietary patterns and gastrointestinal alterations in ASD. Noteworthy findings will contribute to the sparse literature on the association between dietary intervention and neurodevelopmental disorders, and assist with obtaining future funding for higher-level clinical trials involving collaborative research with other medical centers and academic institutions. These initiatives, the investigators believe, are necessary to establish the KD as a novel, safe alternative to effectively treat patients with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2-21 years.
* Primary diagnosis of autism spectrum disorder.
* Parent/legal guardian and child able to read or understand English, and able/willing to provide informed consent/assent.
* Females of childbearing potential must have a negative pregnancy test result and agree to use a medically acceptable method of contraception throughout the entire study period and for 30 days after the last dose of study drug - childbearing potential is defined a girls who are > Tanner stage 2 and urine pregnancy tests are acceptable.

Exclusion Criteria:

* Known cardiac disorder including arrhythmias or hypertension.
* BMI < 3rd%ile.
* Carnitine deficiency (primary).
* Carnitine palmitoyltransferase (CPT) I or II deficiency.
* Carnitine translocase deficiency.
* Beta-oxidation defects - medium-chain acyl dehydrogenase deficiency (MCAD), long-chain acyl dehydrogenase deficiency (LCAD), short-chain acyld dehydrogenase deficiency (SCAD), long-chain 3-hydroxyacyl-coenzyme A (CoA) deficiency, and medium-chain 3-hydroxyacyl-CoA deficiency.
* Pyruvate carboxylase deficiency.
* Porphyria.
* Inability to maintain adequate nutrition.
* Patient or caregiver non-compliance.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 119 (Actual)
Dates: Start 2015-03; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in core symptoms of ASD | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess core autistic symptoms through review/analysis of responses to the following measurement instruments: Autism Diagnostic Observation Schedule - Second Edition (ADOS-2); Asperger Syndrome Diagnostic Scale (ASDS); Childhood Autism Rating Scale (CARS-2); Gilliam Autism Rating Scale (GARS-3); Social Responsiveness Scale - Second Edition (SRS-2); Diagnostic and Statistical Manual IV Text Revision (DSM-IV-TR) and DSM-V ASD criteria; standardized intelligence tests (if available, administered by child's school); and Vanderbilt ADHD Diagnostic Teacher Rating Scale Forms (Vanderbilt).

SECONDARY OUTCOMES:
Change from baseline in the number of medications used for ASD management | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess changes through the review/analysis of self-report and medical record data.
Change from baseline in the dosage of medications used for ASD management | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess changes through the review/analysis of self-report and medical record data.
Change from baseline in the number of lab tests ordered for ASD management | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess changes through the review/analysis of self-report and medical record data.
Change from baseline in the number of emergency room or hospital visits for ASD management | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess changes through review/analysis of self-report and medical record data.
Change from baseline in subject/family satisfaction with the ketogenic diet | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess changes in subject/family satisfaction with the ketogenic diet through review/analysis of responses to a questionnaire.
Change from baseline in biochemical profiles due to the ketogenic diet | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess biochemical profile differences and changes through the analysis of serum and urine ketone levels
Change from baseline in biochemical profiles due to the ketogenic diet | Pre- and post-ketogenic diet intervention (at baseline, and after three and six months on the ketogenic diet)
  Assess biochemical profile differences and changes through the analysis of blood and stool (gut microbiome) specimen samples

OTHER OUTCOMES:
Possible effects of the ketogenic diet | Post-ketogenic diet intervention
  Participants on the ketogenic diet will be followed clinically with standard of care until they are 21 years of age to examine the long-term benefits or risks of the KD.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan W Lee, MD, Principal Investigator — Shriners Hospitals for Children, Honolulu
Locations (1):
- Shriners Hospitals for Children - Honolulu, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stafstrom CE, Rho JM. The ketogenic diet as a treatment paradigm for diverse neurological disorders. Front Pharmacol. 2012 Apr 9;3:59. doi: 10.3389/fphar.2012.00059. eCollection 2012. PMID 22509165
- [Background] Evangeliou A, Vlachonikolis I, Mihailidou H, Spilioti M, Skarpalezou A, Makaronas N, Prokopiou A, Christodoulou P, Liapi-Adamidou G, Helidonis E, Sbyrakis S, Smeitink J. Application of a ketogenic diet in children with autistic behavior: pilot study. J Child Neurol. 2003 Feb;18(2):113-8. doi: 10.1177/08830738030180020501. PMID 12693778
- [Background] Mantis JG, Fritz CL, Marsh J, Heinrichs SC, Seyfried TN. Improvement in motor and exploratory behavior in Rett syndrome mice with restricted ketogenic and standard diets. Epilepsy Behav. 2009 Jun;15(2):133-41. doi: 10.1016/j.yebeh.2009.02.038. Epub 2009 Feb 26. PMID 19249385
- [Background] Ruskin DN, Svedova J, Cote JL, Sandau U, Rho JM, Kawamura M Jr, Boison D, Masino SA. Ketogenic diet improves core symptoms of autism in BTBR mice. PLoS One. 2013 Jun 5;8(6):e65021. doi: 10.1371/journal.pone.0065021. Print 2013. PMID 23755170
- [Background] Niederhofer H. Association of attention-deficit/hyperactivity disorder and celiac disease: a brief report. Prim Care Companion CNS Disord. 2011;13(3):PCC.10br01104. doi: 10.4088/PCC.10br01104. PMID 21977364
- [Background] Cryan JF, Dinan TG. Mind-altering microorganisms: the impact of the gut microbiota on brain and behaviour. Nat Rev Neurosci. 2012 Oct;13(10):701-12. doi: 10.1038/nrn3346. Epub 2012 Sep 12. PMID 22968153
- [Background] Harris SL, Handleman JS. Age and IQ at intake as predictors of placement for young children with autism: a four- to six-year follow-up. J Autism Dev Disord. 2000 Apr;30(2):137-42. doi: 10.1023/a:1005459606120. PMID 10832778
- [Background] Mulle JG, Sharp WG, Cubells JF. The gut microbiome: a new frontier in autism research. Curr Psychiatry Rep. 2013 Feb;15(2):337. doi: 10.1007/s11920-012-0337-0. PMID 23307560
- [Background] Wang Y, Kasper LH. The role of microbiome in central nervous system disorders. Brain Behav Immun. 2014 May;38:1-12. doi: 10.1016/j.bbi.2013.12.015. Epub 2013 Dec 25. PMID 24370461
- [Background] Adams JB, Johansen LJ, Powell LD, Quig D, Rubin RA. Gastrointestinal flora and gastrointestinal status in children with autism--comparisons to typical children and correlation with autism severity. BMC Gastroenterol. 2011 Mar 16;11:22. doi: 10.1186/1471-230X-11-22. PMID 21410934
- [Background] Kang DW, Park JG, Ilhan ZE, Wallstrom G, Labaer J, Adams JB, Krajmalnik-Brown R. Reduced incidence of Prevotella and other fermenters in intestinal microflora of autistic children. PLoS One. 2013 Jul 3;8(7):e68322. doi: 10.1371/journal.pone.0068322. Print 2013. PMID 23844187
- [Background] Ming X, Stein TP, Barnes V, Rhodes N, Guo L. Metabolic perturbance in autism spectrum disorders: a metabolomics study. J Proteome Res. 2012 Dec 7;11(12):5856-62. doi: 10.1021/pr300910n. Epub 2012 Nov 9. PMID 23106572
- [Background] Wang L, Christophersen CT, Sorich MJ, Gerber JP, Angley MT, Conlon MA. Elevated fecal short chain fatty acid and ammonia concentrations in children with autism spectrum disorder. Dig Dis Sci. 2012 Aug;57(8):2096-102. doi: 10.1007/s10620-012-2167-7. Epub 2012 Apr 26. PMID 22535281
- [Background] Wang L, Christophersen CT, Sorich MJ, Gerber JP, Angley MT, Conlon MA. Increased abundance of Sutterella spp. and Ruminococcus torques in feces of children with autism spectrum disorder. Mol Autism. 2013 Nov 4;4(1):42. doi: 10.1186/2040-2392-4-42. PMID 24188502
- [Background] Williams BL, Hornig M, Parekh T, Lipkin WI. Application of novel PCR-based methods for detection, quantitation, and phylogenetic characterization of Sutterella species in intestinal biopsy samples from children with autism and gastrointestinal disturbances. mBio. 2012 Jan 10;3(1):e00261-11. doi: 10.1128/mBio.00261-11. Print 2012. PMID 22233678
- [Background] Yap IK, Angley M, Veselkov KA, Holmes E, Lindon JC, Nicholson JK. Urinary metabolic phenotyping differentiates children with autism from their unaffected siblings and age-matched controls. J Proteome Res. 2010 Jun 4;9(6):2996-3004. doi: 10.1021/pr901188e. PMID 20337404
- [Background] De Angelis M, Piccolo M, Vannini L, Siragusa S, De Giacomo A, Serrazzanetti DI, Cristofori F, Guerzoni ME, Gobbetti M, Francavilla R. Fecal microbiota and metabolome of children with autism and pervasive developmental disorder not otherwise specified. PLoS One. 2013 Oct 9;8(10):e76993. doi: 10.1371/journal.pone.0076993. eCollection 2013. PMID 24130822
- [Background] Hsiao EY, McBride SW, Hsien S, Sharon G, Hyde ER, McCue T, Codelli JA, Chow J, Reisman SE, Petrosino JF, Patterson PH, Mazmanian SK. Microbiota modulate behavioral and physiological abnormalities associated with neurodevelopmental disorders. Cell. 2013 Dec 19;155(7):1451-63. doi: 10.1016/j.cell.2013.11.024. Epub 2013 Dec 5. PMID 24315484
- [Background] Sandler RH, Finegold SM, Bolte ER, Buchanan CP, Maxwell AP, Vaisanen ML, Nelson MN, Wexler HM. Short-term benefit from oral vancomycin treatment of regressive-onset autism. J Child Neurol. 2000 Jul;15(7):429-35. doi: 10.1177/088307380001500701. PMID 10921511
- [Derived] Allan NP, Yamamoto BY, Kunihiro BP, Nunokawa CKL, Rubas NC, Wells RK, Umeda L, Phankitnirundorn K, Torres A, Peres R, Takahashi E, Maunakea AK. Ketogenic Diet Induced Shifts in the Gut Microbiome Associate with Changes to Inflammatory Cytokines and Brain-Related miRNAs in Children with Autism Spectrum Disorder. Nutrients. 2024 May 7;16(10):1401. doi: 10.3390/nu16101401. PMID 38794639